CLINICAL TRIAL: NCT03842319
Title: Impact of MEditerranean Diet, Inflammation and Microbiome on Plaque Vulnerability and Microvascular Dysfunction After an Acute Coronary Syndrome. A Randomized, Controlled, Mechanistic Clinical Trial.
Brief Title: Impact of MEditerranean Diet, Inflammation and Microbiome After an Acute Coronary Syndrome
Acronym: MEDIMACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: Hospital General Universitario Gregorio Marañon (Other); Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other); University of Navarra (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Tel Aviv University (Other); Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CIBER-MEDIMACS
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Atherosclerosis; Mediterranean diet; microbiota; immune system; metabolome; proteome
MeSH Terms: conditions — Acute Coronary Syndrome; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Intervention Group: High intensity Mediterranean diet in secondary prevention after acute coronary syndrome. Control Group: recommendation of a standard of care, standard Mediterranean diet. Duration of the intervention per participant: 12 months. Follow-up period per participant: 12 months.
Who Masked: Investigator
Masking Description: Non-intervention or MedDiet intensive intervention group assignment will be made through an automated system. Each patient will be assigned a patient identification number that should appear on all eCRF pages (electronic "case report"), source documents and laboratory data. All researchers involved in the measurement of data, analysis and allocation of results will be blind. The MedDiet intensive intervention will be blind to the evaluation of the endpoints (the research team in charge of the measurement, analysis and awarding of the results will be blind). The samples will be coded and anonymously analyzed by each research team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): In patients allocated to the control group, the currently used Spanish Mediterranean diet will be recommended as part of a standard high-quality secondary prevention program, where the patient is invited to participate in a single 45 minute nutritional educational group session. Interventions: Microbiota analysis, Immunological analysis, Proteome analysis, Metabolome analysis, Clinical evaluation
  Interventions: Other: Microbiota analysis; Other: Immunological analysis; Other: Proteome analysis; Other: Metabolome analysis; Other: Clinical evaluation; Other: Diet evaluation
- High-intensity MedDiet (Experimental): Patients allocated to the interventional group will be individually evaluated by a dietitian and will participate in dedicated individual and group sessions at baseline, and at 3, 6, 9 and 12 months. In the interventional group, a personalized MedDiet will assess chemical and nutritional composition and total energy intake will be adapted to participant's weight, age, and requirements, and the dietitian's tailored advice to his/her individual needs. A 14-item dietary screen for adherence to the Mediterranean diet will be used to personalize the intervention and negotiate dietary changes. Furthermore, free virgin olive oil, recipes, shopping list and designed weekly menus will be provided to maximize the differences between groups. Interventions: MedDiet, Microbiota analysis, Immunological analysis, Proteome analysis, Metabolome analysis, Clinical evaluation, Diet evaluation
  Interventions: Other: Microbiota analysis; Other: Immunological analysis; Other: Proteome analysis; Other: Metabolome analysis; Other: Clinical evaluation; Other: Diet evaluation; Other: MedDiet

INTERVENTIONS:
Other: Microbiota analysis — From the feces and oral cavity samples, the DNA of the microbiota will be extracted using specific extraction kits and the microbiome will be analyzed through the study of 16S ribosomal RNA amplicons.
Other: Immunological analysis — A study of immunological cell populations, inmunogenetics and cytokines will be carried out from fresh blood samples using antibody panels and flow cytometry
Other: Proteome analysis — A study of host and microbiota proteome will be carried out from samples using mass spectrometry
Other: Metabolome analysis — A study of host and microbiota metabolome will be carried out from samples using MS-based as well as NMR-based methods
Other: Clinical evaluation — Clinical evaluation including hemostasis and biochemical studies
Other: Diet evaluation — Biochemical analysis and questionaries for diet adherence and exercise registration
Other: MedDiet — The high-intensity Mediterranean diet will include the promotion of the following: a) abundant use of olive oil (>40 g/d) for cooking and dressing dishes; b) consumption of >2 daily servings of vegetables; c) >2-3 daily serving of fresh fruits; d) >3 weekly servings of legumes; e) >3 weekly servings of fish or seafood; f) >1 weekly serving of nuts or seeds; g) select white meats instead of red meats or processed meats; and h) cook regularly with tomato, garlic and onion adding or no other aromatic herbs, and dress vegetables, pasta, rice and other dishes with tomato, garlic and onion adding or no other aromatic herbs. Two main meals per day should be eaten (seated at a table, lasting more than 20 minutes). A recommendation to drink a glass of wine per day during meals is given. Limited consumption is advised for cured ham, red meat, chocolate, cured or fatty cheeses
  Arms: High-intensity MedDiet

SUMMARY:
In the MEDIMACS project, the investigators will use a randomized clinical-trial design to address the effects of mediterranean diet on atherosclerotic plaque vulnerability and coronary endothelial function in order to decipher complex interplays between diet, microbiome, immunological and metabolic responses and coronary atherosclerosis. The investigators will focus on patients after an episode of acute coronary syndrome and use state-of-the-art techniques to address atherosclerotic plaque composition and coronary endothelial function. A number of different -omic approaches will be used to address effector pathways. The insights provided by this study will allow identifying potential new dietary, microbiota and/or metabolic targets for the treatment of atherosclerosis

DETAILED DESCRIPTION:
Coronary atherosclerosis is a leading cause of mortality and disability worldwide. Continuous efforts are needed to improve secondary prevention and understand the mechanism underlying disease progression. Based on primary prevention trials, a potential benefit of the Mediterranean diet after an acute coronary syndrome can be anticipated. The integrated microbiome-mediated/ immunologic and metabolic pathways by which the Mediterranean diet modifies cardiovascular risk remain mostly unknown. Intestinal and oral dysbiosis is involved in the pathogenesis of atherosclerosis and microbiome dynamics may account for some of the observed benefits of Mediterranean diet. The first objective of the trial is to evaluate the effects of a well-controlled Mediterranean diet intervention on atherosclerotic plaque vulnerability and coronary endothelial dysfunction after an episode of acute coronary syndrome. The second objective is to decipher the interplays among diet, microbiota, immunity and metabolism responsible for the observed effects. The investigators propose a randomized mechanistic clinical trial, using state-of-the-art efficacy read-outs. The multidisciplinary consortium includes highly experienced cardiologists, nutritionists and experts in translational research in immunology, microbiomics, genomics, proteomics, metabolomics and metagenomics. This study will provide valuable insights to identify potential microbiome therapeutic targets for coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiac catheterization for an acute coronary syndrome.
* At least 1 non-causal lesion in a coronary segment with a stenosis diameter between 40-70% that will not be submitted to intervention during the revascularization procedure.
* Disposition and possibility to modify the diet.
* With the ability to track and answer questionnaires.
* Signature of informed consent for the study

Exclusion Criteria:

* TIMI score <3 in the injury
* Reference lesion with diameter <2.0 mm
* LV ejection fraction (EF) less than 45%.
* Active systemic infection
* Active periodontal disease
* Chronic inflammatory disease
* Active treatment with corticosteroids or immunomodulators
* Renal insufficiency with glomerular filtration less than 30 mL / min
* Severe hepatic insufficiency (liver cirrhosis in Child B or C stages).
* Comorbidity with life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Fibrous cap thickness change | 12 months
  Change in the thickness of the fibrous layer of the atheroma plaque in the non-culprit vessel measured by optical coherence tomography at 12 months.

SECONDARY OUTCOMES:
Endothelial dysfunction | 12 months
  Vascular endothelial function measured using a Doppler pressure guidewire
Intestinal microbiota composition changes | 12 months
  Changes from baseline in intestinal microbiota will be analysed using the 16S rRNA target gene sequencing approach at 3 months, 6 months, 9 months and 12 months
Oral microbiota composition changes | 12 months
  Changes from baseline in oral microbiota will be analysed using the 16S rRNA target gene sequencing approach at 3 months, 6 months, 9 months and 12 months
Adaptive immune system status changes | 12 months
  Changes from baseline of adaptive immune cell lineages will be assessed dynamically using high performance cytometry at 3 months, 6 months, 9 months and 12 months
Innate immune system status changes | 12 months
  Changes from baseline of innate immune cell lineages will be assessed dynamically using high performance cytometry at 3 months, 6 months, 9 months and 12 months
Blood protein profiling changes | 12 months
  Changes from baseline of host protein-profiles from collected plasma samples will be analyzed for detection of biomarkers at 3 months, 6 months, 9 months and 12 months
Faecal protein profiling changes | 12 months
  Changes from baseline of host protein-profiles from collected faces samples will be analyzed for detection of biomarkers at 3 months, 6 months, 9 months and 12 months
Urine metabolome profiling changes | 12 months
  Changes from baseline of host metabolome profiles in urine will be analyzed using mass-spectrometry-based at 3 months, 6 months, 9 months and 12 months
Blood metabolome profiling changes | 12 months
  Changes from baseline of host metabolome profiles in blood will be analyzed using mass-spectrometry-based at 3 months, 6 months, 9 months and 12 months
Faecal metabolome profiling changes | 12 months
  Changes from baseline of metabolome profiles in faecal samples will be analyzed using mass-spectrometry-based at 3 months, 6 months, 9 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Fernández-Avilés, Professor, Principal Investigator — CIBER, HGUGM
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The Consortium Partners involved in data creation and analysis agrees to follow the FAIR data management principles of Findability, Accessibility, Interoperability and Reusability. The Project Management Committee will decide what type and format of data to be stored in the collective database and what type and format of data will be available publicly (as an open-access to research data), as well as how data will be curated and preserved after the end of the project. Sequences, genotypes and protein and immune profiles would be organized and indexed in metadata files following a unique code of assignment that will be submitted for releasing to public database repositories such as GenBank, Gene Expression Omnibus and ClinicalTrials. The International Standards for Genomes and Metagenomes will be followed

REFERENCES:
- [Derived] Fernandez AI, Bermejo J, Yotti R, Martinez-Gonzalez MA, Mira A, Gophna U, Karlsson R, Al-Daccak R, Martin-Demiguel I, Gutierrez-Ibanes E, Charron D, Fernandez-Aviles F; MEDIMACS research team. The impact of Mediterranean diet on coronary plaque vulnerability, microvascular function, inflammation and microbiome after an acute coronary syndrome: study protocol for the MEDIMACS randomized, controlled, mechanistic clinical trial. Trials. 2021 Nov 12;22(1):795. doi: 10.1186/s13063-021-05746-z. PMID 34772433